CLINICAL TRIAL: NCT06546254
Title: A Double-blind Randomized Controlled Trial of 1% Lidocaine Paracervical Block for Endometrial Biopsy
Brief Title: 1% Lidocaine Paracervical Block for Endometrial Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Mara Sobel, Prinicipal Investigator (Dr.), Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: REB 23-0078-A
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Biopsy
Keywords: lidocaine
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: The proposed study is a double-blind randomized controlled trial. Participants will be recruited from Mount Sinai Hospital outpatient gynecology clinics. Recruitment, consent, randomization, procedure, and post-procedure survey will occur during the same visit. Each participant will be randomly assigned to one of two arms:
  Each participant will be randomly assigned to one of two arms:
  1. intervention (paracervical block - 10 mL 1% lidocaine with epinephrine)
  2. control (gently tapping the cervicovaginal junction with a capped needle)
  The primary outcome will be a global pain score, which will be patient-reported by the 100 mm Visual Analogue Scale (VAS) following the procedure.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigators will employ a two provider system to ensure a double-blinded set-up. The first provider (Provider A) will open the allocation envelopes without the presence of the participant or second provider (Provider B).
  Provider A will then enter the patient's room and introduce themselves. Provider A will place the speculum, and administer either the intervention or control and then leave the room after injection-related bleeding has stopped. After 3 minutes, the second provider (Provider B) will enter the room to place the tenaculum and perform the endometrial biopsy and will be unaware of the participant's treatment arm.
  A standardized script will be used with all participants: "You may or not may feel a poke."
  Both lidocaine and the control are odorless and clear, minimizing the risk of unblinding. All data will remain blinded until data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1% lidocaine paracervical injection (Experimental): 10 cc 1% lidocaine with epinephrine paracervical injection
  Interventions: Drug: Lidocaine 1% Injectable Solution
- control (Sham Comparator): gently tapping the cervicovaginal junction with a capped needle
  Interventions: Other: Capped needle

INTERVENTIONS:
Drug: Lidocaine 1% Injectable Solution — 10 cc 1% lidocaine paracervical injection
  Arms: 1% lidocaine paracervical injection
Other: Capped needle — Tapping the cervicovaginal junction with a capped needle
  Arms: control

SUMMARY:
The objective of this study is to to determine whether 1% lidocaine paracervical block reduces pain during endometrial biopsy in comparison to no intervention.

The proposed study is a double-blind randomized controlled trial (RCT).

Each participant will be randomly assigned to one of two arms:

1. intervention (paracervical block - 10 mL 1% lidocaine with epinephrine)
2. control (gently tapping the cervicovaginal junction with a capped needle)

The primary outcome will be a global pain score, which will be patient-reported by the 100 mm Visual Analogue Scale (VAS) following the procedure.

ELIGIBILITY:
Inclusion Criteria

* Any participant > or = age 18 years old presenting for an endometrial biopsy
* All parities of patients are eligible
* English speaking participants only

Exclusion Criteria

* Use of pain medication that is not an NSAID or acetaminophen (e.g. opioids, benzos) within past 24 hours
* Confirmed pregnancy
* Any diagnosed chronic pain syndromes (eg. fibromyalgia, vaginismus, interstitial cystitis)
* Contraindication to lidocaine
* Misoprostol administration within 24 hours
* Previous unsuccessful office attempt at endometrial biopsy by the same practitioner (note of clarification: previous unsuccessful biopsy attempt by a different practitioner will still be eligible)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Global pain score | Immediately after the completion of the procedure
  100 mm Visual Analogue Scale (VAS), minimum value 0 (no pain at all) and maximum value 100 (worst pain imaginable)

SECONDARY OUTCOMES:
Pain scores during procedure | During the procedure
  Pain rating on scale of 0 - 10 at the following time points: baseline, after injection/control, placement of tenaculum, endometrial biopsy completion, 1-minute post-biopsy
Immediate complications of endometrial biopsy and/or intervention/control | Immediately after the completion of the procedure
  Provider reported
Difficulty for provider to complete the biopsy | Immediately after the completion of the procedure
  Provider reported on Likert scale, minimum 1 (least difficult) and maximum 5 (most difficult)
Length of time for analgesia | During procedure
  Stopwatch
Length of time for endometrial biopsy completion | During procedure
  Stopwatch
Number of passes with biopsy pipelle to collect sufficient tissue | Immediately after the completion of the procedure
  Provider reported
Amount of tissue obtained: scant, minimal, adequate | Immediately after the completion of the procedure
  Provider reported
Patient satisfaction | Immediately after the completion of the procedure
  Survey

CONTACTS AND LOCATIONS:
Locations (1):
- OPG, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No